CLINICAL TRIAL: NCT03368846
Title: An Open Label, Single-dose, Single-period Study Designed to Assess the Mass Balance Recovery, Metabolite Profile and Metabolite Identification of [14C]-Varlitinib in Healthy Male Subjects
Brief Title: Open, Single-dose/-Period Study to Assess Mass Balance Recovery, Metabolite Profile/Identification of 14C-Varlitinib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ASLAN Pharmaceuticals (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ASLAN001-018
Record Dates: First submitted 2017-11-22; First posted 2017-12-11 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]-Varlitinib (Experimental)
  Interventions: Drug: Varlitinib

INTERVENTIONS:
Drug: Varlitinib — [14C]-Varlitinib

SUMMARY:
This is a single-centre, open-label, non-randomised, single oral dose study in healthy male subjects. It is planned to enrol a single cohort of 6 healthy male subjects to ensure data in 4 evaluable subjects.

Each subject will receive a single administration of 120 mg [14C] varlitinib oral suspension containing not more than (NMT) 2.9 MBq (79 µCi), in the fed state.

DETAILED DESCRIPTION:
Subjects will be screened for eligibility to participate in the study up to 28 days before dosing. Subjects will be admitted to the clinical unit on the evening prior to IMP administration (Day 1) and will fast overnight for a minimum of 8 h. Subjects will be dosed on the morning of Day 1 following a light breakfast, and will remain resident in the clinic until up to 240 h after dosing (Day 11). It is planned that subjects will be released as a group when all subjects have achieved a mass balance cumulative recovery of >90%, or if <1% of the dose administered has been collected in urine and faeces within 2 separate, consecutive 24 h periods. In this case, collection of all samples (blood, urine and faeces) will cease and the subjects will undergo discharge assessments. If this criterion has not been met by all subjects on Day 11, the residency period may be extended by a further 48 h maximum (up to Day 13). If the criterion is still not met by Day 13, or if additional residency is not considered appropriate or necessary, then home collections of urine and/or faeces may be requested at the discretion of the investigator for individual subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males of non-Asian descent
2. Aged 30 to 65 years
3. Body mass index of 18.0 to 35.0 kg/m2 or, if outside the range, considered not clinically significant by the investigator
4. Must be willing and able to communicate and participate in the whole study
5. Must provide written informed consent
6. Must agree to use an adequate method of contraception (as defined in Section 9.4)
7. Must have regular bowel movements (ie, average stool production of ≥1 and ≤3 stools per day)
8. Subject is considered healthy on the basis of medical history, physical examination, ECG, vital signs and clinical laboratory assessments.

Exclusion Criteria:

1. Subjects who have received any IMP in a clinical research study within the previous 3 months
2. Subjects who are study site employees, or immediate family members of a study site or sponsor employee
3. Subjects with pregnant partners
4. Subjects who have previously been enrolled in this study
5. History of any drug or alcohol abuse in the past 2 years
6. Regular alcohol consumption in males >21 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine)
7. Current smokers and those who have smoked within the last 12 months. A breath carbon monoxide reading of greater than 10 ppm at screening and admission
8. Users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months
9. Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 1999, shall participate in the study
10. Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator at screening
11. Clinically significant abnormal biochemistry, haematology or urinalysis as judged by the investigator (laboratory parameters are listed in Appendix 1)
12. Neutrophil count <1.8 x109/L at screening
13. ALT and AST >1.25 x upper limit of normal range at screening
14. QT interval corrected for heart rate using Fridericia's formula (QTcF) > 450 msec at screening
15. Positive drugs of abuse test result (drugs of abuse tests are listed in Appendix 1)
16. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
17. Evidence of renal impairment at screening, as indicated by an estimated creatinine clearance (CLcr) of <80 mL/min using the Cockcroft-Gault equation
18. History of clinically relevant cardiovascular, renal, hepatic, chronic respiratory or Gl disease, neurological or psychiatric disorder, as judged by the investigator
19. History of clinically relevant dermatological disease (eg eczema, psoriasis, drug rashes) or the presence of dermatological conditions at screening (eg acne, eczema, dermatitis etc)
20. Subjects with a history of cholecystectomy or gall stones
21. Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
22. Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hayfever is allowed unless it is active
23. Donation or loss of greater than 400 mL of blood within the previous 3 months
24. Subjects who are taking, or have taken, any prescribed or over-the-counter drug or herbal remedies in the 14 days before IMP administration; with the exception of 4 g per day paracetamol [see Section 11.4]). Further exceptions may apply on a case by case basis, if considered not to interfere with the objectives of the study, as agreed by the PI and sponsor's medical monitor.
25. Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-11-23 (Actual); Primary Completion 2017-12-06 (Actual); Study Completion 2017-12-14 (Actual)

PRIMARY OUTCOMES:
Mass balance recovery after a single oral dose of [14C] varlitinib | Assessments will be made up to 13 days postdose
  Mass balance recovery of [14C] varlitinib recovered in urine, faeces, and all excreta
Metabolite profiling and structural identification of metabolites in plasma, urine and faeces | Assessments will be made up to 13 days postdose
  Identification of the chemical structure of metabolites

SECONDARY OUTCOMES:
Routes and rates of elimination of [14C] varlitinib | Assessments will be made up to 13 days postdose
  Amount [14C] varlitinib excreted for urine and faeces
Determination of the chemical structure of the "major" metabolites of [14C] varlitinib | Assessments will be made up to 13 days postdose
  Identification of the chemical structure of each metabolite accounting for greater than 10%
Evaluation of whole blood:plasma concentration ratios for total radioactivity | Assessments will be made up to 13 days postdose
PK of total radioactivity and varlitinib in plasma following a single oral dose of [14C] varlitinib | Assessments will be made up to 13 days postdose
  Peak Plasma Concentration (Cmax)
PK of total radioactivity and varlitinib in plasma following a single oral dose of [14C] varlitinib | Assessments will be made up to 13 days postdose
  Area under the plasma concentration versus time curve (AUC)
PK of total radioactivity and varlitinib in plasma following a single oral dose of [14C] varlitinib | Assessments will be made up to 13 days postdose
  Half life
PK of total radioactivity and varlitinib in plasma following a single oral dose of [14C] varlitinib | Assessments will be made up to 13 days postdose
  The time from dosing at which Cmax was apparent
Collect additional information on the safety and tolerability of varlitinib | Assessments will be made up to 13 days postdose
  Number of participants with abnormal laboratory values and/or adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Clinical Ltd, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No